CLINICAL TRIAL: NCT01780025
Title: Clinical Trial on Objective Measures in Implantable Hearing Devices for Subjects With Mixed Hearing Loss.
Brief Title: Objective Measures in Implantable Hearing Devices
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Sponsor
Other Study IDs: S53530
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2023-01-27 (Actual); Status verified 2013-01

CONDITIONS: Mixed Hearing Loss
Keywords: Hearing; Thresholds; Coupling to the inner ear
MeSH Terms: conditions — Hearing Loss, Mixed Conductive-Sensorineural | interventions — Evoked Potentials, Auditory; Hearing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mixed hearing loss
  Interventions: Behavioral: Auditory evoked potentials and audiometry; Behavioral: Auditory evoked potentials

INTERVENTIONS:
Behavioral: Auditory evoked potentials and audiometry
Behavioral: Auditory evoked potentials — Different protocols for audiometry and auditory evoked potentials

SUMMARY:
The purpose of this study is to measure objectively the coupling from direct acoustic cochlear stimulation to the inner ear with a non-invasive technique of auditory evoked potentials.

DETAILED DESCRIPTION:
A new technique, called Direct Acoustic Cochlear Stimulation, has very recently been introduced to restore hearing in patients with severe hearing loss due to the immobility of a small ossicle in the middle ear, the stapes. A piston-like prosthesis, which is placed up into the inner ear, is connected to an implantable mechanical stimulator, named DACS. Unfortunately, as with other active middle ear implants, until now the correct function of this technique cannot be checked during the surgery, leading to a possibly variable outcome of hearing. In this project, the objective auditory evoked potentials, like Auditory Steady-State Response (ASSR), will be used to measure the efficacy of this method of inner ear stimulation. This highly innovative, non-invasive research will provide valuable insight in a new promising way of inner ear stimulation and may give a unique possibility to measure the correct connection from an implantable hearing device to the inner ear.

ELIGIBILITY:
Inclusion Criteria:

* adults
* mixed hearing loss

Exclusion Criteria:

* children

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mixed hearing loss
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2012-04; Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
auditory evoked potentials | 1 - 3 - 6 months

SECONDARY OUTCOMES:
speech audiometry | 3 and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium